CLINICAL TRIAL: NCT00080548
Title: Timing of Voluntary Movement in Patients With Schizophrenia Using EEG and Surface EMG
Brief Title: Timing of Voluntary Movement in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040151; 04-N-0151
Record Dates: First submitted 2004-04-07; First posted 2004-04-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-06

CONDITIONS: Schizophrenia
Keywords: Bereitschafts Potential; Timing of Volition; Somatic Passivity Phenomenon; Conscious Will; Libet's Clock; Schizophrenia; Healthy Volunteer; HV
MeSH Terms: conditions — Schizophrenia

SUMMARY:
This study will examine and compare how the brain controls the timing of movement in healthy volunteers and in people with schizophrenia. Previous experiments have shown that when people are asked to look at a clock and report the time they first decide to make a movement, they report times later than the first brain waves associated with movement appear. When they are asked to report the time they first initiate the movement, they report times before the muscles actually begin to move. The study may help determine how the sense of willing and initiating an action is altered in schizophrenic patients, and how people may feel more or less "in control" of their movements.

Normal volunteers and patients with schizophrenia between 18 and 65 years of age may be eligible for this study. Control subjects must not have any neurological or psychological disorders, and schizophrenia patients must not have any other neurological disorders.

All participants will have a medical history, physical examination, and a test to determine their level of attention. Schizophrenia patients will be interviewed about their symptoms and complete psychiatric rating scales. In addition, all participants will undergo the following procedures:

Electric shock

Participants look at a clock on a computer screen whose hands revolves around the clock fast. While they look at the clock, they are given small, non-painful electric shocks and are asked to say when they receive the shocks, according to the clock. The shocks are repeated 40 times.

Arm movement

Participants are asked to lift their arm up off a table repeatedly, at random times, while they look at the computer clock. This exercise is repeated a total of 80 times. Of these 80 times, participants are asked 10 times in a row to say the time they first had the desire to move their arm, and then 10 times in a row the time they first felt that they were moving their arm.

Electroencephalography (EEG) and Electromyography (EMG)

Participants undergo EEG and EMG during the electric shock and arm movement experiments to measure electrical activity of the brain (EEG) and of the muscles (EMG). For EEG, electrodes (small metal discs) are placed on the scalp with a cap, paste, or glue-like substance and the brain waves are recorded. For EMG, electrodes are taped to the skin over the muscle.

DETAILED DESCRIPTION:
Objectives

The purpose of this study is to determine how the subjective sense of willing and initiating an action is altered in schizophrenic patients. One proposed explanation for characteristic symptoms of schizophrenia ("passivity phenomena") is a defect in the forward model of movement that the brain receives as the motor signal is generated. We propose to examine this forward model using Libet's paradigm, in which normal subjects gave evidence for a forward model in their anticipatory reports of initiation of movement. We intend to determine the times associated with willing (W), initiating (M), and electroencephalographic/electromyographic (EEG/EMG) measures of movement.

Study Population

We intend to study adult patients with a Diagnostic and Statistical Manual of Mental Disorders diagnosis of schizophrenia. These patients provide a unique population for this study because they often do not have the sense that they direct their own movement or author their own thoughts (passivity phenomena). Studies have shown that schizophrenics have movement-related cortical potentials on EEG, but it is not known when the subjective sense of initiating movement occurs for these patients. As the order of mental events in time has been shown to contribute to the sense of agency, it is important to know how the timing of voluntary movement is altered in schizophrenia.

Design

We will ask patients to look at a fast-rotating clock on a computer screen and note when their movements were willed, instigated by an external agent if they have such delusions, and were initiated. Patients will also report the time of a somatosensory stimulus. Surface EMG will determine the time of actual movement, and EEG will record brain potentials associated with movement. Eligible patients with schizophrenia and passivity phenomena will be recruited from the Clinical Brain Disorders Branch, NIMH.

Outcome Measures

The primary outcome measure of this study is the absence of time W in some schizophrenics, the latency of W in other schizophrenics compared to normal subjects, and the latency of M in schizophrenics compared to normals. Any effect of medication status or symptoms on performance in the study will be considered exploratory data.

ELIGIBILITY:
* INCLUSION CRITERIA:

SCHIZOPHRENIC PATIENTS:

Experimental subjects will be patients with DSM-IV diagnosis of schizophrenia who have volunteered to participate in the clinical research unit of the Clinical Brain Disorders Branch, NIMH. In addition, outpatients with DSM-IV diagnosis of schizophrenia who participate in outpatient research through the CBDB will be included. All patients will have received the diagnosis of schizophrenia by means of the Structured Clinical Interview for DSM-IV (SCID) with three psychiatrists reaching a consensus diagnosis. Patients on the clinical research unit must meet rigorous criteria in order to participate in research. Exclusionary criteria include history of traumatic brain injury, known comorbid neurological disorders, including epilepsy, history of drug and alcohol abuse, etc. All patients will have undergone a comprehensive battery of neuropsychological tests, including Wide Range Achievement Test- Reading (often to be a good indicator of premorbid intelligence), a short version of Wechsler Adult Intelligence Scale (WAIS-R), Wechsler Memory Scales (WMS-R), Trails A and B, tests of attention and executive function, including the continuous performance test (CPT), Wisconsin Card Sort (WISC), the N-Back test of working memory. Patients with psychiatric diseases other than schizophrenia that are not currently active and symptomatic will be included.

All patients in the study will have schizophrenia. However, at the time of testing, patients will be administered clinical rating scales (i.e., Brief Psychotic Rating Scale (BPRS), appropriate sections of the SCID and the Yale Hallucination Phenomenology Assessment (YHPA)) to determine the presence of passivity phenomena.

NORMAL VOLUNTEERS:

Twenty-six normal controls will be included; controls will be screened in the NINDS Movement Disorders Outpatient Clinic, and will have neurological and physical examinations. They will be asked to abstain from alcohol for 24 hours before the study. All subjects participating in the studies will have a valid Clinical Center Medical Record Number.

ALL SUBJECTS:

All subjects will be between the ages of 18 and 65. Subjects may be male or female.

EXCLUSION CRITERIA:

Patients younger than 18 years old or older than 65 years old will be excluded from the study.

A. Patients with neurological disorders will be excluded. Patients with psychiatric disorders other than schizophrenia who are experiencing an active phase of their disorder will be excluded.

B. Patients with a history of significant medical disorders requiring chronic treatment with other drugs, which affect the central nervous system and cannot be stopped will be excluded.

C. Patients not capable of giving an informed consent will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-04-06; Study Completion 2009-01-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blakemore SJ, Smith J, Steel R, Johnstone CE, Frith CD. The perception of self-produced sensory stimuli in patients with auditory hallucinations and passivity experiences: evidence for a breakdown in self-monitoring. Psychol Med. 2000 Sep;30(5):1131-9. doi: 10.1017/s0033291799002676. PMID 12027049
- [Background] Chapman LJ, Chapman JP. The measurement of differential deficit. J Psychiatr Res. 1978;14(1-4):303-11. doi: 10.1016/0022-3956(78)90034-1. No abstract available. PMID 722633
- [Background] Frith CD, Done DJ. Experiences of alien control in schizophrenia reflect a disorder in the central monitoring of action. Psychol Med. 1989 May;19(2):359-63. doi: 10.1017/s003329170001240x. PMID 2762440